CLINICAL TRIAL: NCT05274503
Title: Serum Interleukine 6 as a Predictor of Outcome in Mechanically Ventilated Patients With Covid 19
Brief Title: Interleukine 6 as a Predictor of Outcome in Mechanically Ventilated Patients With Covid 19
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Mokhtar Ahmed, lecturer of anesthesia and intensive care, Sohag University
Other Study IDs: soh-Med-22-1-27
Record Dates: First submitted 2022-03-09; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Mechanical Ventilation Duration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Serum IL-6 levels will be determined by enzyme-linked immunosorbent assay according to the manufacturer's instructions and the normal range is <10 pg/mL , Patients' medical records will be carefully reviewed and analyzed. Patient data regarding demographics, comorbidities, signs and symptoms, laboratory results and complications will be collected. The occurrence of complications will be confirmed according to the following criteria: acute respiratory distress syndrome (ARDS) defined according to the Berlin definition

ELIGIBILITY:
Inclusion Criteria:

* •Age: more than 20 years.

  * Gender: both males and females will be included.
  * Mechanically Ventilated patients.
  * COVID 19 confirmed diagnosis

Exclusion Criteria:

* •Immunocompromised patients.

  * Oxygen saturation more than 95% without ventilation.
  * Malignancy.
  * Patients refuse to be enrolled in the study.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients more than 20 years old, covid positive, mechanically ventilated
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
detection of acute respiratory distress syndrome | 2 weeks
  hypoxia, incresed plateau pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Faculty of Medicine, Sohag, Egypt